CLINICAL TRIAL: NCT04810949
Title: Effect of Vitamin D Supplementation on the Development of Respiratory Infections (COVID-19) in Health Personnel at Hospital Clínica NOVA With Serum Values> 20ng / ml
Brief Title: Vitamine D3 Supplementation in Patients With Serum Values +/- 20ng/ml
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: patients enrolled got vaccinated vs COVID-19 and Influenza
Sponsor: Hospital Clinica Nova (Other)
Responsible Party: Principal Investigator, Maria Elena Romero Ibarguengoitia, Principal Investigator/Research Director, Hospital Clinica Nova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vitamina D NOVA
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Influenza A; Influenza B; H1N1 Influenza
MeSH Terms: conditions — COVID-19; Orthomyxoviridae Infections | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- serum vitamin D levels >20ng/ml (Group 1) (Experimental): Patients with serum vitamin D levels >20ng/ml that will receive Vitamin D supplementation
  Interventions: Dietary Supplement: Vitamine D3 supplementation
- serum vitamin D levels >20ng/ml ( Group 2) (Experimental): Patients with vitamin D levels >20ng/ml that will receive diet and hygiene measures
  Interventions: Dietary Supplement: Diet and sun exposure
- serum vitamin D3 levels < 20ng/ml (Group3) (Other): Patients with Vitamin D levels<20ng/ml will receive vitamin D3 supplementation according to primary care discresion
  Interventions: Dietary Supplement: Vitamine D3 supplementation

INTERVENTIONS:
Dietary Supplement: Vitamine D3 supplementation — 1. The supplementation treatment will consist of prescribing vitamin D3 consumption of 4000 U 13 single dose tablets each month (52,000 IU).
  Arms: serum vitamin D levels >20ng/ml (Group 1); serum vitamin D3 levels < 20ng/ml (Group3)
Dietary Supplement: Diet and sun exposure — 2. Hygienic-dietary recommendations will consist of 2 steps
  1. Sun exposure at least 10 minutes a day from 10: 00-6: 00 pm
  2. Consumption of foods rich in vitamin D: milk, fish, almonds, mushrooms
  Arms: serum vitamin D levels >20ng/ml ( Group 2)

SUMMARY:
Scarce information exists in relation to the effect of supplementation of Vitamin D3 in SARS-COV-2 infection, H1N1, and A, B Influenza when 25-hydroxyvitamin levels are between 20-100ng/ml. This study will evaluate the effect of supplementation of vitamin D3 vs. dietary-hygiene measures in SARS-COV-2 , H1N1, A, B Influenza infection rate in patients with serum 25-hydroxyvitamin D3 levels >20ng/ml.

A comparative randomized study that will evaluate the effect of a monthly supplementation with 52000 units of Vitamine D3 during three months vs hygienic-dietary measures in the development of respiratory infections such as COVID-19, H1N1, A, B Influenza during 6 months of follow-up in health workers from a hospital in Northern Mexico with serum vitamin D values +/- 20ng/ml. Also, patients that during screening have 25-hydroxyvitamin D3 levels <20 ng/ml will receive vitamin D supplementation according to primary care discretion for three months and will be followed for 6 months and infection rate will be analyzed and compared.

DETAILED DESCRIPTION:
COVID-19 is an infectious disease caused by the newly discovered coronavirus SARS-CoV-2, with a clinical spectrum from asymptomatic infection to critical and fatal illnesses. Influenza H1N1, A, and B have also been the most frequent etiologies of respiratory tract infection that are usually affected during the winter season before COVID-19 pandemic.

There is controversy against Vitamin D3 supplementation in the prevention of respiratory tract infections. A previous meta-analysis has demonstrated an association between vitamin D3 levels <20mg/dl and a higher risk of infection. There is less information in relation to the effect of supplementation when vitamin levels are between 20-100ng/ml and the prevention of infection.

The rationale of this study will be to find a relationship between vitamin D3 supplementation and the incidence of SARS-CoV-2 or Influenza H1N1, A, or B infection through a prospective study. Vitamin D3 could have a role in innate and adaptive immunity that could help prevent this disease. The target population will be health workers with a high risk of SARS-COV-2 or influenza infection with vitamin D > 20 ng/ml.

The primary aim is to evaluate the effect of vitamin D3 supplementation vs. dietary-hygiene measures in developing SARS-COV-2 infection, Influenza H1N1, A or B in patients with serum 25-hydroxyvitamin D3 >20 ng/ml.

A secondary aim will be to compare a group of hospital workers with serum 25-hydroxyvitamin D3 < 20 ng/ml that could or not have been supplemented with Vitamin D3.

Hypothesis primary aim: There will be no difference in the development of respiratory infections (COVID-19, H1N1 Influenza, A, B influenza) in health personnel with serum levels of vitamin D equal or greater than 20ng / ml when they receive supplementation vs treatment based on hygienic-dietary measures (diet and sun exposure), in a 6-month follow-up.

The hypothesis of secondary aim: the infection rate of COVID-19, and H1N1, A or B influenza will be higher in the group of vitamin D3 <20ng/ml than the patients with levels between 20-100ng/ml

A comparative quasi-experimental study that will evaluate the effect of 2 treatments in health workers of Hospital Clínica Nova with serum vitamin D values > 20ng / ml. The study will be conducted per The Code of Ethics of the World Medical Association (Declaration of Helsinki) for humans experiments and also will be approved by the local IRB from Universidad de Monterrey.

1. Supplementation with 52,000 units of vitamin D3 monthly
2. Hygienic-dietary measures: sun exposure 10 minutes a day plus recommendation of consumption of foods rich in vitamin D.

Baseline serum levels will be assessed, and monthly follow-up will be given regarding the development of symptoms suggestive of respiratory tract infection. The monitoring of serum levels of vitamin D will be every 3 months.

Efficacy endpoint: During the follow-up period, the most effective treatment will develop a lower respiratory tract infection rate ( COVID-19 and/or H1N1, A or B Influenza ).

Procedures:

1. Serum levels of vitamin D (25-hydroxyvitamin D) will be measured in all medical personnel working at Hospital Clínica Nova.
2. Patients with Vitamin D3<20ng/ml will be supplemented by primary care physician
3. Treatment group will be randomized to patients with vitamin D3 levels >20ngml.
4. Serum vitamin D levels will be monitored every 3 months
5. Monthly follow-up will be given through the endocrinology consultation on the development of respiratory symptoms

Secondary endpoint: Personnel with vitamin D levels <20ng/ml will be sent to a primary care physician for treatment by the doctor's discretion and will be followed for the same period of time in order to evaluate COVID-19 and H1N1, A or B Influenza infection rate.

The relative risks that could be presented in the different groups are an increase of Vitamin D serum levels > 100ng /ml in the G1 and a reduction of vitamin D serum levels < 20ng/ml in G2. To reduce the risk, serum vitamin D3 levels will be monitored every three months.

Statistical analysis Two researchers will review the quality control of the database and anonymized it. Normality assumption will be evaluated with the Shapiro Wilk test and frequency histograms. Descriptive statistics such as mean, the standard deviation for quantitative variables, frequencies, and percentages for categorical variables, will be computed. Chi-square tests and ANOVA will be used to compare the categorical and quantitative data between groups. Kaplan-Mayer, Log-rank, and Cox regression were used for the analysis of SARS-COV-2 development.

Missing data were handled by complete case analysis. For simple randomization, we will use a random number generation with binomial distribution with a probability of 50%.

The sample size will be of a finite population as it will include all health personnel who work at Hospital Clínica Nova.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Both genders
* Absence of infection by COVID-19, influenza H1N1, influenza A or B at the time of measurement of serum vitamin D levels.
* Absence of infection at any site of bacterial, fungal or other origins
* Health worker at Hospital Clínica Nova.

Patient Exclusion Criteria for both arms:

* Serum Vitamin D levels> 100ng / ml
* Previous consumption of supplements containing Vitamin D3
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Covid-19 Infection with Vitamin D3 > 20ng/ml | 6 months
  Evaluate the number of patients that get infected by COVID-19 during study period with vitamin D3 levels >20ng/ml that receive supplementation or diet and hygiene measures
Number of participants with Influenza H1N1 infection with Vitamin D3 > 20ng/ml | 6 months
  Evaluate the number of patients that get infected by H1N1 infection with vitamin D3 levels +/- 20ng/ml that receive supplementation or diet or hygiene measures
Number of participants with Influenza A infection with Vitamin D3 > 20ng/ml | 6 months
  Evaluate the number of patients that get infected by Influenza A with vitamin D3 levels +/- 20ng/ml that receive supplementation or diet or hygiene measures
Number of participants with Influenza B infection with Vitamin D3 > 20ng/ml | 6 months
  Evaluate the number of patietns that get infected by Influenza B with vitamin D3 levels +/- 20ng/ml that receive supplementation or diet or hygiene measures

SECONDARY OUTCOMES:
Number of participants with Covid-19 Infection with Vitamin D3 < 20ng/ml | 6 months
  Evaluate the number of patients that get infected by COVID-19 during study period with vitamin D3 levels <20ng/ml that receive supplementation according to primary care physician
Number of participants with H1N1 infection Infection with Vitamin D3 < 20ng/ml | 6 months
  Evaluate the number of patients that get infected by H1N1 during study period with vitamin D3 levels <20ng/ml that receive supplementation according to primary care physician prescription
Number of participants with influenza A Infection with Vitamin D3 < 20ng/ml | 6 months
  Evaluate the number of patients that get infected by Influenza A during study period with vitamin D3 levels <20ng/ml that receive supplementation according to primary care physician prescription
Number of participants with influenza B Infection with Vitamin D3 < 20ng/ml | 6 months
  Evaluate the number of patients that get infected by Influenza B during study period with vitamin D3 levels <20ng/ml that receive supplementation according to primary care physician prescription

CONTACTS AND LOCATIONS:
Overall Officials: Arnulfo Gonzalez-Cantu, MD, Principal Investigator — Hospital Clinica Nova
Locations (1):
- Hospital Clinica Nova de Monterrey, San Nicolás de los Garza, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: during one year after the publication of the results
Access Criteria: contacting corresponding author

REFERENCES:
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Spiteri G, Fielding J, Diercke M, Campese C, Enouf V, Gaymard A, Bella A, Sognamiglio P, Sierra Moros MJ, Riutort AN, Demina YV, Mahieu R, Broas M, Bengner M, Buda S, Schilling J, Filleul L, Lepoutre A, Saura C, Mailles A, Levy-Bruhl D, Coignard B, Bernard-Stoecklin S, Behillil S, van der Werf S, Valette M, Lina B, Riccardo F, Nicastri E, Casas I, Larrauri A, Salom Castell M, Pozo F, Maksyutov RA, Martin C, Van Ranst M, Bossuyt N, Siira L, Sane J, Tegmark-Wisell K, Palmerus M, Broberg EK, Beaute J, Jorgensen P, Bundle N, Pereyaslov D, Adlhoch C, Pukkila J, Pebody R, Olsen S, Ciancio BC. First cases of coronavirus disease 2019 (COVID-19) in the WHO European Region, 24 January to 21 February 2020. Euro Surveill. 2020 Mar;25(9):2000178. doi: 10.2807/1560-7917.ES.2020.25.9.2000178. PMID 32156327
- [Background] Griffin G, Hewison M, Hopkin J, Kenny RA, Quinton R, Rhodes J, Subramanian S, Thickett D. Perspective: Vitamin D supplementation prevents rickets and acute respiratory infections when given as daily maintenance but not as intermittent bolus: implications for COVID-19. Clin Med (Lond). 2021 Mar;21(2):e144-e149. doi: 10.7861/clinmed.2021-0035. Epub 2021 Feb 16. PMID 33593830
- [Background] Dzopalic T, Bozic-Nedeljkovic B, Jurisic V. The role of vitamin A and vitamin D in modulation of the immune response with a focus on innate lymphoid cells. Cent Eur J Immunol. 2021;46(2):264-269. doi: 10.5114/ceji.2021.103540. Epub 2021 Aug 7. PMID 34764797
- [Background] Bilezikian JP, Bikle D, Hewison M, Lazaretti-Castro M, Formenti AM, Gupta A, Madhavan MV, Nair N, Babalyan V, Hutchings N, Napoli N, Accili D, Binkley N, Landry DW, Giustina A. MECHANISMS IN ENDOCRINOLOGY: Vitamin D and COVID-19. Eur J Endocrinol. 2020 Nov;183(5):R133-R147. doi: 10.1530/EJE-20-0665. PMID 32755992
- [Background] Ilie PC, Stefanescu S, Smith L. The role of vitamin D in the prevention of coronavirus disease 2019 infection and mortality. Aging Clin Exp Res. 2020 Jul;32(7):1195-1198. doi: 10.1007/s40520-020-01570-8. Epub 2020 May 6. PMID 32377965
- [Background] Oristrell J, Oliva JC, Casado E, Subirana I, Dominguez D, Toloba A, Balado A, Grau M. Vitamin D supplementation and COVID-19 risk: a population-based, cohort study. J Endocrinol Invest. 2022 Jan;45(1):167-179. doi: 10.1007/s40618-021-01639-9. Epub 2021 Jul 17. PMID 34273098
- [Background] Dror AA, Morozov N, Daoud A, Namir Y, Yakir O, Shachar Y, Lifshitz M, Segal E, Fisher L, Mizrachi M, Eisenbach N, Rayan D, Gruber M, Bashkin A, Kaykov E, Barhoum M, Edelstein M, Sela E. Pre-infection 25-hydroxyvitamin D3 levels and association with severity of COVID-19 illness. PLoS One. 2022 Feb 3;17(2):e0263069. doi: 10.1371/journal.pone.0263069. eCollection 2022. PMID 35113901
- [Background] Demir M, Demir F, Aygun H. Vitamin D deficiency is associated with COVID-19 positivity and severity of the disease. J Med Virol. 2021 May;93(5):2992-2999. doi: 10.1002/jmv.26832. Epub 2021 Feb 9. PMID 33512007
- [Background] Chiodini I, Gatti D, Soranna D, Merlotti D, Mingiano C, Fassio A, Adami G, Falchetti A, Eller-Vainicher C, Rossini M, Persani L, Zambon A, Gennari L. Vitamin D Status and SARS-CoV-2 Infection and COVID-19 Clinical Outcomes. Front Public Health. 2021 Dec 22;9:736665. doi: 10.3389/fpubh.2021.736665. eCollection 2021. PMID 35004568
- [Background] Loucera C, Pena-Chilet M, Esteban-Medina M, Munoyerro-Muniz D, Villegas R, Lopez-Miranda J, Rodriguez-Bano J, Tunez I, Bouillon R, Dopazo J, Quesada Gomez JM. Real world evidence of calcifediol or vitamin D prescription and mortality rate of COVID-19 in a retrospective cohort of hospitalized Andalusian patients. Sci Rep. 2021 Dec 3;11(1):23380. doi: 10.1038/s41598-021-02701-5. PMID 34862422
- [Background] Quesada-Gomez JM, Entrenas-Castillo M, Bouillon R. Vitamin D receptor stimulation to reduce acute respiratory distress syndrome (ARDS) in patients with coronavirus SARS-CoV-2 infections: Revised Ms SBMB 2020_166. J Steroid Biochem Mol Biol. 2020 Sep;202:105719. doi: 10.1016/j.jsbmb.2020.105719. Epub 2020 Jun 11. PMID 32535032
- [Background] Martinez-Moreno JM, Herencia C, Montes de Oca A, Munoz-Castaneda JR, Rodriguez-Ortiz ME, Diaz-Tocados JM, Peralbo-Santaella E, Camargo A, Canalejo A, Rodriguez M, Velasco-Gimena F, Almaden Y. Vitamin D modulates tissue factor and protease-activated receptor 2 expression in vascular smooth muscle cells. FASEB J. 2016 Mar;30(3):1367-76. doi: 10.1096/fj.15-272872. Epub 2015 Dec 23. PMID 26700731
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368